CLINICAL TRIAL: NCT01183884
Title: 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid for Consolidation of Second or Greater Remission of High-Risk Neuroblastoma: A Phase II Study
Brief Title: 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid for Consolidation of Second or Greater Remission of High-Risk Neuroblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low participant accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-160
Record Dates: First submitted 2010-08-16; First posted 2010-08-18 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2018-09

CONDITIONS: Neuroblastoma
Keywords: GM-CSF; MAB 3F8; RETINOIC ACID (CIS-9 & 13); 09-160
MeSH Terms: conditions — Neuroblastoma | interventions — Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid (Experimental): This phase II, open-label, single arm trial assesses the anti-NB activity of high-dose 3F8 (80 mg/m2/day), which is used in cycles 1-2, with return to standard 3F8 dosage (20 mg/m2/day) in subsequent cycles. Clinical results will be compared to those in the predecessor trials which used only the standard 3F8 dosage. Starting with A(6), patients no longer receive high-dose 3F8 but receive only standard dose 3F8 (20 mg/m2/day) for all cycles.
  Interventions: Biological: 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid

INTERVENTIONS:
Biological: 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid — 3F8 (80 mg/m2/day), which is used in cycles 1-2, with return to standard 3F8 dosage (20 mg/m2/day) in subsequent cycles .Clinical results will be compared to those in the predecessor trials which used only the standard 3F8 dosage.
  Starting with A(6), patients no longer receive high-dose 3F8 but receive only standard dose 3F8 (20 mg/m2/day) for all cycles. The patients are in > or = to 2nd CR/VGPR and at high risk for additional relapse. Real-time quantitative RT-PCR63-65 will be used to assess MRD in BM. 13-cis-retinoic acid is started after cycle 2.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, the combination of 3F8 and GM-CSF has on the patient and the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NB as defined by a) histopathology (confirmed by the MSKCC Department of Pathology), or b) BM metastases or MIBG-avid lesion(s) plus high urine catecholamine levels.
* High-risk NB as defined by risk-related treatment guidelines1 and the International NB Staging System,89 i.e., stage 4 with (any age) or without (> or = to 18 months of age) MYCN amplification, MYCN-amplified stage 2 or stage 3 (any age), or MYCN-amplified stage 4S.
* The patients are in >2nd CR/VGPR, including no measurable MIBG-avid soft tissue tumor assessable for response.
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Creatinine > 3.0 mg/dL
* ALT, AST and Alkaline Phosphatase > 5.0 times the upper limit of normal
* Bilirubin > 3.0 mg/dL
* Patients with grade 3 or higher toxicities (using the CTCAE v34.0) related to cardiac, neurological, pulmonary or gastrointestinal function as determined by physical exam. Patients must have normal blood pressure for age.
* Progressive disease
* History of allergy to mouse proteins
* Active life-threatening infection.
* Human anti-mouse antibody (HAMA) titer >1000 Elisa units/ml.
* Inability to comply with protocol requirements.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-08; Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Kushner BH, Modak S, Basu EM, Roberts SS, Kramer K, Cheung NK. Posterior reversible encephalopathy syndrome in neuroblastoma patients receiving anti-GD2 3F8 monoclonal antibody. Cancer. 2013 Aug 1;119(15):2789-95. doi: 10.1002/cncr.28137. Epub 2013 Apr 30. PMID 23633099
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid
Started | 46
Completed | 8
Not Completed | 38
Not completed — Progressive Disease | 26
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Other Complicating Disease | 3
Not completed — Not Treated | 1
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Arm/Group | 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 6 [1 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 41
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Assess the Impact of High-dose 3F8/GM-CSF on Relapse-free Survival
Description: in patients in second or greater complete or very good partial remission, but at high risk of additional relapse.
Time Frame: 2 years
Population: Data not collected
Arm/Group | 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid
Number analyzed (Participants) | 0

2. Secondary Outcome: Apply Real-time Quantitative RT-PCR to Test the Hypothesis That the Minimal Residual Disease Content of Bone Marrow
Description: after the first treatments with 3F8/GMCSF has significant prognostic impact on relapse-free survival.
Time Frame: 2 years
Population: Data not collected
Arm/Group | 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid
Number analyzed (Participants) | 0

3. Secondary Outcome: Monitor Safety of the High-dose Antibody Treatment
Description: to assure no side-effects or noxious sequelae develop or emerge that were not seen in the prior phase I study.
Time Frame: 2 years
Population: Data not collected
Arm/Group | 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Only mortality data collected, Serious and Other Adverse Events not monitored/assessed.
Arm/Group | 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid
All-Cause Mortality (participants affected / at risk) | 24/46
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT01183884/Prot_SAP_000.pdf